CLINICAL TRIAL: NCT01848210
Title: Evaluation of Efficacy and Safety of the Fixed-dose Combination of Coumarin and Troxerutin (Venalot®) Versus Placebo in the Symptomatic Treatment of Chronic Venous Insufficiency - VENACT
Brief Title: Efficacy and Safety of Coumarin and Troxerutin in the Symptomatic Treatment of Chronic Venous Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VN01/12; U1111-1141-7277 (Other: World Health Organization); 15030313.0.1001.5470 (Other: CAAE)
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Venous Insufficiency
Keywords: Drug therapy
MeSH Terms: interventions — coumarin; troxerutin; Venalot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coumarin 30 mg + Troxerutin 180 mg (Experimental): Coumarin 30 mg, troxerutin 180 mg fixed-dose combination tablets, orally, three times daily for up to 16 weeks.
  Interventions: Drug: Coumarin/troxerutin
- Placebo (Placebo Comparator): Coumarin + troxerutin placebo-matching tablets, orally, three times daily for up to 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coumarin/troxerutin — Coumarin + troxerutin fixed-dose combination tablets
  Other Names: Venalot®
  Arms: Coumarin 30 mg + Troxerutin 180 mg
Drug: Placebo — Coumarin + troxerutin placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the fixed-dose combination of coumarin and troxerutin versus placebo in the symptomatic treatment of chronic venous insufficiency.

DETAILED DESCRIPTION:
The drug being tested in this study is the fixed-dose combination of coumarin and troxerutin called Venalot®. Venalot is being tested to treat the symptoms of chronic venous insufficiency. This study will look at symptom relief in people who take Venalot®.

The study will enroll approximately 808 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Combination coumarin + troxerutin extended release tablets
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take two tablets three times a day throughout the study.

This multi-centre trial will be conducted in Brazil. The overall time to participate in this study is up to 18 weeks. Participants will make 6 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Consent of subject or legal representative
2. Men or women of any ethnicity, aged between 18 and 75 years, and body mass index (BMI) equal or less than 40.
3. Is able to use properly the medication according to protocol.
4. Has chronic venous insufficiency in the reference leg with the clinical classification C3, or C4a orC4b or C5, provided that in two last situations the present lipodermatosclerosis does not compromise more than 1/3 portion of the leg immersed or immersible in the plethysmometer.
5. Has stable edema (in a steady state), equivalent to a variation lower than or equal to 10% in partial volume of the reference leg between the screening visit and the randomization visit, and present for at least 6 months.
6. Scoring in "Severity Score of Local Complaints" equal to or higher than 5 total points.
7. Women who are using an effective (at the discretion of the investigator), but not hormonal, birth control method (not hormonal intrauterine device (IUD), surgical sterilization, among others), or who are postmenopausal, in addition to condom use (mandatory).

Exclusion Criteria:

1. Has chronic venous insufficiency classified as C1, C2 in the reference leg or C6 in any leg.
2. Has chronic venous insufficiency C4b or C5 in the reference leg, with lipodermatosclerosis present in more than 1/3 portion of the leg immersed in the plethysmometer.
3. Has unstable edema, equivalent to variation of more than 10% of partial volume in the reference leg between the screening visit and randomization visit, prior to start of treatment.
4. Has venous obstruction and/or deep vein thrombosis (DVT) and/or presence of phlebitis in lower limbs during the last 3 (three) months.
5. Has developed deep vein insufficiency during the last 3 (three) months.
6. Has other diseases that may interfere in the findings of the study such as: lymphedema, thrombosis, clotting disorders, edema of lower limbs due to right-sided heart failure, arterial obstruction of lower limbs and other conditions that, at medical discretion, are relevant to exclusion, particularly symptoms which are similar to the symptomatology of chronic venous insufficiency.
7. Has a history of surgery at the venous system or sclerotherapy or who received any treatment for chronic venous insufficiency during the last 03 months, whether it was by drug, elastic stocking, laser, or surgery.
8. Has used previously Venalot® and had no benefits with the treatment.
9. Has a previous history of known or suspected allergy or intolerance to any of the ingredients of the medicinal product under investigation.
10. Has any clinical finding (history and physical examination) that is interpreted by the physician-investigator as a risk to participant's participation in the study.
11. Has known serious systemic disease, according to the medical and/or laboratory history.
12. Has history of a known liver disease such as hepatitis A, hepatitis B, or C.
13. Has changed at least one lab parameters: aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyltransferase (gamma-GT), or alkaline phosphatase 2.5 times above the upper limit of normal range; hemoglobin less than 10 g/dL; clearance of creatinine estimative equal or above 60mL/min/1.73 m^2; platelets below 90,000/mL; and total bilirubin and fractions 1.5 times above the normal values.
14. Has been using diuretics for a period less than or equal to 6 months due to any disease (hypertension, renal failure, or other).
15. Has serious chronic liver or kidney disease, according to the medical and/or laboratory history.
16. Has uncontrolled blood hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg) at randomization or clinical hypertensive urgency.
17. Has a previous history of diabetes mellitus on use of insulin.
18. Has received treatment with immunosuppressive drugs, including systemic corticosteroids within 30 days before the start of study (randomization visit), or who are receiving immunosuppressive treatments, or who have known congenital or acquired immunodeficiency.
19. Has malignant neoplasms, from any etiology, or who are receiving any type of anticancer treatment, unless when properly treated and with no evidence of recurrence during the last five years. Non-melanoma skin cancer is not an exclusion criterion.
20. Is unable to understand the guidelines specified in this protocol or who cannot attend all the study visits.
21. Has a previous history of alcoholism, drug abuse, psychological or emotional problems in the last 5 years that can invalidate the Informed Consent Form or restrain participant's ability to comply with the requirements of the protocol.
22. Pregnant or breastfeeding women, or those who have the potential to become pregnant and are not using an appropriate contraceptive method.
23. Women who are using hormonal contraceptives or hormone replacement treatment, including phytoestrogens, within the last 3 months.
24. Took part in clinical trials during the last year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- [Derived] Martinez-Zapata MJ, Vernooij RW, Simancas-Racines D, Uriona Tuma SM, Stein AT, Moreno Carriles RMM, Vargas E, Bonfill Cosp X. Phlebotonics for venous insufficiency. Cochrane Database Syst Rev. 2020 Nov 3;11(11):CD003229. doi: 10.1002/14651858.CD003229.pub4. PMID 33141449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Brazil from 28 May 2013 to 29 September 2015.
Pre-assignment Details: Participants with a diagnosis of chronic venous insufficiency were enrolled equally in 1 of 2 treatment groups, three times a day coumarin 30 mg and troxerutin 180 mg fixed-dose combination tablets or matching placebo.
Groups:
- Coumarin + Troxerutin: Coumarin 30 mg, troxerutin 180 mg fixed-dose combination tablets, orally, three times daily for up to 16 weeks.
Period: Overall Study
Arm/Group | Coumarin + Troxerutin | Placebo
Started | 411 | 418
Safety Population-Received Study Drug | 394 | 398
Intent-to-Treat (ITT) Population | 383 | 388
Per Protocol Population | 222 | 245
Completed | 323 | 340
Not Completed | 88 | 78
Not completed — Informed Consent Form Withdrawal | 28 | 24
Not completed — Lost to Follow-up | 24 | 12
Not completed — Protocol Violation | 3 | 5
Not completed — Use of Forbidden Drugs | 9 | 10
Not completed — Impedition Condition | 5 | 9
Not completed — Adverse Event | 7 | 9
Not completed — Discontinuation Criterion | 5 | 7
Not completed — Hypesensitivity | 1 | 0
Not completed — Hepatic Function Alteration | 4 | 0
Not completed — Chronic Venous Insufficiency Course | 1 | 2
Not completed — Administrative | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population included all eligible participants who received study drug and had at least one efficacy assessment at Visit 1 (28 ± 5 days after start of treatment).
Groups:
- Total: Total of all reporting groups
Arm/Group | Coumarin + Troxerutin | Placebo | Total
Number analyzed (Participants) | 383 | 388 | 771
Age, Continuous [Mean (Full Range); unit: years] | 55.95 [20.00 to 75.00] | 55.81 [20.00 to 75.00] | 55.88 [20.00 to 75.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337 | 351 | 688
  Male | 46 | 37 | 83
Race/Ethnicity, Customized [Number; unit: participants]
  White | 221 | 240 | 461
  Black | 48 | 55 | 103
  Brown | 110 | 86 | 196
  Asian | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  Brazil | 383 | 388 | 771
Height [Mean (Full Range); unit: meters] | 1.58 [1.35 to 1.87] | 1.59 [1.43 to 1.89] | 1.59 [1.35 to 1.89]
Weight [Mean (Full Range); unit: kg] | 74.40 [45.00 to 133.00] | 73.38 [45.00 to 114.00] | 73.89 [45.00 to 133.00]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/cm^2] | 29.76 [19.91 to 39.96] | 29.14 [19.63 to 39.86] | 29.45 [19.63 to 39.96]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change (Reduction) From Baseline in Volume of Reference Leg at Week 16
Description: Change in the partial volume of legs will be measured using a water plethysmometer. The volume of water (at 34 ± 0.2 °C) displaced after limb immersion is collected in an empty plastic Beaker which has been previously weighed (scale tare). The equilibrium/stability will be estimated using the absolute difference between measures of volume obtained at the Week 16 visit and Baseline to determine the reduction in edema.
Time Frame: Baseline and Week 16
Population: Participants from the ITT population, all eligible participants who received study drug and had at least one efficacy assessment at Visit 1 (28 ± 5 days after start of treatment), with data available for analysis.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Coumarin + Troxerutin | Placebo
Number analyzed (Participants) | 333 | 347
milliliters (mL) | 1.13 (93.67) | 5.78 (107.26)
Statistical Analysis 1: Comparison: Coumarin + Troxerutin vs Placebo; Test type: Superiority or Other; p = 0.531, Regression, Linear; Mean Difference (Final Values) = -4.65, 95% CI 2-sided [-19.81 to 10.51]

2. Secondary Outcome: Change (Reduction) From Baseline in Local Complaint Severity
Description: Local Complaint Severity will be assessed using the Severity Score of Local Complaints that comprises 8 items: 1=tired legs, 2=heavy legs, 3= feeling of tension, 4=feeling of swelling, 5=aching legs, 6=tingling, 7=itching, 8=burning of soles of the feet.
  Each item is classified with a Likert-type scale of 5 levels, where 0=absent, 1=low, 2=medium, 3=high, 4=very high.
  A total score is calculated from the sum of the scores of all the 8 items and ranges from 0 (complaints absent) to 32 (very high severity).
Time Frame: Baseline and Week 16
Population: ITT population, all participants who received study drug and had at least one efficacy assessment at Visit 1 (28 ± 5 days after start of treatment). Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coumarin + Troxerutin | Placebo
Number analyzed (Participants) | 382 | 388
score on a scale | 10.83 (6.70) | 10.45 (6.97)

3. Secondary Outcome: Overall Assessment by the Investigator
Description: The investigator recorded their impression of the overall clinical picture at the end of the treatment period (Week 16), taking into account the clinical picture compared with the Baseline visit. Data is reported for the percentage of participants in each of the following assessment categories: worsening, unchanged, discreet improvement or accentuated improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Coumarin + Troxerutin | Placebo
Number analyzed (Participants) | 340 | 356
percentage of participants
  Worsening | 0.6 | 0.8
  Unchanged | 11.2 | 14.3
  Discreet improvement | 25.3 | 24.4
  Accentuated improvement | 62.9 | 60.4

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse events are any unwanted medical occurrences in an individual taking part in a clinical study who is receiving a pharmaceutical product. The adverse event does not have necessarily a causal relationship with the treatment. In this definition, any adverse or unwanted signals and symptoms, or findings that appear from the start or that deteriorate during the clinical study are also included, i.e. any intercurrent diseases (recently diagnosed concomitant diseases or symptoms), accidents and clinically relevant changes in clinical laboratory values.
Time Frame: Baseline to Week 16
Population: Safety Population included all randomized participants who received study drug and had a least one post-Baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Coumarin + Troxerutin | Placebo
Number analyzed (Participants) | 394 | 398
participants | 131 | 120

ADVERSE EVENTS:
Time Frame: From the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator documented any occurrence of adverse events. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of relation to study treatment. Safety Population: all randomized participants who received study drug and had a least one post-Baseline safety assessment.
Arm/Group | Coumarin + Troxerutin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/394 | 2/398
Other Adverse Events (participants affected / at risk) | 115/394 | 81/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coumarin + Troxerutin (N=394) | Placebo (N=398)
Varicose vein operation (Surgical and medical procedures) | 1 | 2
Phlebectomy (Surgical and medical procedures) | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Coumarin + Troxerutin (N=394) | Placebo (N=398)
Abdominal pain upper (Gastrointestinal disorders) | 12 | 6
Gastritis (Gastrointestinal disorders) | 7 | 7
Nausea (Gastrointestinal disorders) | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 5 | 1
Influenza like illness (General disorders) | 4 | 3
Influenza (Infections and infestations) | 4 | 15
Tonsillitis (Infections and infestations) | 7 | 5
Urinary tract infection (Infections and infestations) | 6 | 6
Gamma-glutamyltransferase increased (Investigations) | 7 | 3
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Obesity (Metabolism and nutrition disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Headache (Nervous system disorders) | 16 | 10
Dizziness (Nervous system disorders) | 4 | 3
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 4
Hypertension not otherwise specified (NOS) (Vascular disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 30 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results.